CLINICAL TRIAL: NCT00450047
Title: Study on the Efficacy of Speed-Feedback Therapy for Elderly People With Dementia: a Randomized Controlled Trial
Brief Title: Study on the Efficacy of Speed-Feedback Therapy for Elderly People With Dementia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hiroshima University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0662
Record Dates: First submitted 2007-03-20; First posted 2007-03-21 (Estimated); Last update posted 2007-03-21 (Estimated); Status verified 2007-03

CONDITIONS: Dementia
Keywords: cognitive impairment, ergometer, speed-feedback therapy
MeSH Terms: conditions — Dementia; Cognitive Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Speed-feedback therapy system with a bicycle ergometer
Device: Ergometer at conventional settings

SUMMARY:
The purpose of this study is to verify the efficacy of speed-feedback therapy in improving the cognitive function of elderly people with dementia by a randomized controlled trial, and to demonstrate how that affects ADL and QOL.

DETAILED DESCRIPTION:
Dementia is a syndrome caused by diseases of the cerebral parenchyma, and it is a state in which cognitive functions, including attention, memory, thinking, comprehension, judgment, and computation, are diminished. Because of the mental symptoms, problem behaviors, and decreased activities of daily living (ADL) it is also recognized as a major social problem. However, rehabilitation of elderly people with dementia is still at the trial-and-error stage, and establishing a method of rehabilitation is an urgent task. In 2004, the authors devised and created a training method that integrates exercise therapy with feedback therapy to treat the cognitive dysfunction of elderly people with dementia. To do so the authors introduced speed-feedback therapy with a bicycle ergometer as a feedback therapy intervention. The results of a preliminary study of the efficacy of this method in improving cognitive dysfunction in 17 elderly persons with dementia showed improvement in cognitive dysfunction, and their attentiveness also improved, suggesting that the impaired attentiveness may have improved in response to treatment by this method and, as a result, have led to improvement of cognitive dysfunction. However, it became clear that it would be necessary to further improve and develop the system, and to demonstrate its efficacy in a controlled trial and verify associations between improvement of cognitive dysfunction and improvement of the ADL of dementia patients and their quality of life (QOL).

ELIGIBILITY:
Inclusion Criteria:

1. 65 years of age or older
2. Diagnosed with dementia by a physician
3. Mini-Mental State Examination score of 23 points or less
4. Capable of participating at least once a week for 6 weeks in succession

Exclusion Criteria:

1. Management of a medical risk required
2. Impaired ability to pedal the ergometer because of an orthopedic or surgical disease of the lower extremities or central nerve paralysis
3. Never having been on a bicycle, and incapable of pedaling well

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 120
Dates: Start 2005-09; Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
score on a scale of cognitive function immediately after completion of the 6-week intervention and 1 month after completion of the intervention

SECONDARY OUTCOMES:
attentiveness score immediately after completion of the intervention, and score on an ADL scale and a QOL scale immediately after completion of the intervention and 1 month after completion of the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Hitoshi Okamura, MD, PhD, Study Director — Graduate School of Health Sciences, Hiroshima University